CLINICAL TRIAL: NCT02502539
Title: Cellular and Molecular Adaptations to Exercise-induced Inflammatory Response in Children With Autoimmune Diseases
Acronym: AJI-APA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0234; 2015-A00607-42 (Registry Identifier: 2015-A00607-42)
Record Dates: First submitted 2015-05-29; First posted 2015-07-20 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Juvenile idiopathic arthritis; Physical exercise; Pro-anti-inflammatory balance; Interleukins; miRNA; Calgranulins
MeSH Terms: conditions — Arthritis, Juvenile; Motor Activity

ARMS (1):
- autoimmune disease (Experimental): to identify the mechanisms through which physical activity is liable to mediate inflammatory balance in autoimmune disease settings, and specifically in JIA patients.
  Interventions: Procedure: Controlled physical activity

INTERVENTIONS:
Procedure: Controlled physical activity

SUMMARY:
Juvenile idiopathic arthritis (JIA) is a chronic disease characterized by persistent joint inflammation. The immune system disruption that leads to overproduction of pro-inflammatory cytokines (TNF-α, IL-1, IL-6) is a cascade of events on different levels-some molecular, some cellular, and some systemic. Our objective is to identify the mechanisms through which physical activity is liable to mediate inflammatory balance in autoimmune disease settings, and specifically in JIA patients.

DETAILED DESCRIPTION:
Feasibility study

ELIGIBILITY:
Inclusion Criteria:

* Children between 8 and 12 years
* Tanner stage < T2
* polyarthritis, oligoarthritis and ERA sub-type of JIA
* Stable disease during 3 months before starting study

Exclusion Criteria:

* Infection
* Fever
* Anti-IL6 treatment
* More than 6h per week of physical activity
* Systemic corticosteroid treatment during the 3 months before starting study
* Systemic JIA
* JIA not mastered by treatments
* Other autoimmunity or auto-inflammatory diseases
* Participation in another clinical research protocol

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-10 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Percent change | AT DAY 1
  Percent change, before and after a controlled session of physical activity session, of serum and secretion kinetics of IL-6 and its soluble receptors (sIL- 6R and sgp130)

SECONDARY OUTCOMES:
pain (VAS) | at day 1
  to assess slipping quality
locomotors function (CHAQ) | at day 1
  to assess slipping quality
swelling of knee | at day 1
  to assess slipping quality
rate of miRNA | at day 1
  to assess slipping quality
plasma level of melatonin | at day 1
  to assess slipping quality
sitfness of knee | at day 1
  to assess slipping quality

CONTACTS AND LOCATIONS:
Overall Officials: Etienne MERLIN, Principal Investigator — CHU ESTAING
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France